CLINICAL TRIAL: NCT06961045
Title: Computer - Guided Inferior Alveolar Nerve Lateralization With Simultaneous Prosthetic Driven Implant Placement
Brief Title: Computer - Guided Inferior Alveolar Nerve Lateralization With Simultaneous Prosthetic Driven Implant Placement Will be Performed on 10 Surgical Sides (Mandibular Quadrants) to Evaluate the Postoperative Neurosensory Disturbances Following Guided Inferior Alveolar Nerve Lateralization
Acronym: IANL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: AYMAN M. ARAKEEP, MSc, PhD researcher (Other)
Responsible Party: Sponsor-Investigator, AYMAN M. ARAKEEP, MSc, PhD researcher, Assistant Lecturer of Oral and Maxillofacial surgery, Tanta University
Organization: Tanta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS 4-24 2184
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Neurosensory Function of Inferior Alveolar Nerve
Keywords: Inferior Alveolar Nerve Lateraliztion; Computer Assisted; Clinical neurosensory Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main single arm for the clinical trial (Other)
  Interventions: Procedure: Guided Inferior Alveolar Nerve Lateralization with Simultaneous Implant Placement

INTERVENTIONS:
Procedure: Guided Inferior Alveolar Nerve Lateralization with Simultaneous Implant Placement — All patients will be operated on under general anesthesia. A para-crestal incision will be done and a mucoperiosteal flap will be reflected exposing the alveolar ridge and the buccal cortex. The surgical guide will be fitted and fixed in place and the outline of the window will be drawn by the aid of the surgical guide using the piezotome then the guide will be removed. Once the osteotomy is completed the bone window will be mobilized for exposure of the neurovascular bundle. The diamond tips will be used for removal of any remaining bone around the nerve. The neurovascular bundle will be dissected and retracted properly. a surgical guide will be inserted for implant osteotomy. The bone block which was removed for the buccal window will be crushed to be particulates and will be mixed with autologous fibrin glue for preparation of sticky bone, the sticky bone will be packed gently in the window area around the neurovascular bundle then will be covered by platelet rich fibrin.

SUMMARY:
The aim of this clinical trial is to primarily evaluate the postoperative neurosensory disturbances following guided inferior alveolar nerve lateralization with simultaneous implant placement in 10 surgical sides (mandibular quadrants distal to the mental foramen) either in males or females with age range from 30 to 75 years. The main questions it aims to answer are:

1. Will the postoperative neurosensory disturbances after the surgical intervention fade out and if not, will it be annoying to the patient?
2. Can we consider inferior alveolar nerve lateralization efficient substitute to short implants?
3. will the inserted implants going to be properly ossteointegrated at the site of osteotomy for lateralization?

ELIGIBILITY:
Inclusion Criteria:

* Atrophic mandibular ridges distal to the mental foramen with residual alveolar bone height ≤ 8 mm above the IAN.
* The width of the alveolar ridge ≥ 6 mm, 3mm down from the alveolar crest.

Exclusion Criteria:

* All patients suffering from any systemic disease that may contraindicate implant surgery or affect bone healing and osseointegration of implant.
* Previous history of bone augmentation or implant placement in the site planned for nerve lateralization.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
clinical neurosensory testing of the inferior alveolar nerve function | Postoperatively 1 week, 1 month, 3 months, 6 months
  We will use the light touch test and sensitivity mapping by applying moderated pressure with a periodontal probe to depress the skin by 1-2 mm while the patients will be seated comfortably in a quiet room with their eyes closed throughout the procedures. We will show the hypo aesthetic area as a graphic to illustrate its extension. We will choose this technique because it selects the dysfunction of rapidly adapting long myelinated fibers, which are 90% of the fibers of the IAN.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Egypt, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
every necessary individual participant data required for any publication will be shared
Supporting Information: Study Protocol, SAP, ICF